CLINICAL TRIAL: NCT07166731
Title: High Coverage CARotid Stenting vs. Medical Management Alone to Prevent EmboliSm From symptomaTic Non-stenotic cARotid Disease (SyNC) - CARESTAR
Brief Title: High Coverage CARotid Stenting vs. Medical Management Alone to Prevent EmboliSm From symptomaTic Non-stenotic cARotid Disease (SyNC)
Acronym: CARESTAR
Status: Not yet recruiting | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CARESTAR Study
Record Dates: First submitted 2025-08-07; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Carotid Artery Disease; Symptomatic Carotid Artery Stenosis; Carotid Artery Stenting; Carotid Plaque Imaging; Embolic Stroke of Undetermined Source; Carotid Artery Thrombosis
Keywords: SyNC; Carotid artery disease; carotid artery stenting; symptomatic non-stenotic carotid artery disease; carotid artery stenosis; symptomatic carotid artery stenosis
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Artery Thrombosis; Carotid Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular Treatment Group: This group will be both given medical treatment according to standard clinical routine and treated by carotid artery stenting with the high coverage carotid stent (CARESTO® heal, Acandis® Pforzheim)
- Best medical treatment group: This group will be given medical treatment according to standard clinical routine

SUMMARY:
Goal is to analyse the clinical safety and efficacy of the CARESTO® heal Stent within standard clinical routine for the treatment of patients with symptomatic non-stenotic carotid disease (SyNC) and with high-risk plaque features for stroke recurrence compared to medical treatment alone with respect to the mid- and long-term clinical outcomes.

DETAILED DESCRIPTION:
The purpose of the CARESTAR study is to analyse the clinical safety and efficacy of the CARESTO® heal Stent within standard clinical routine for the treatment of patients with symptomatic non-stenotic carotid disease (SyNC) <50% and with high-risk plaque features for stroke recurrence compared to the medical treatment group and with respect to the mid- and long-term clinical outcomes. By randomly assigning participants to the two treatment arms, the aim is to generate bias-free and reliable data that can provide information on the optimal treatment approach in this patient group. Despite advances in medical therapy and endovascular treatment, the optimal treatment strategy for low-grade vulnerable plaques remains unclear. There is therefore an urgent need to evaluate the efficacy and safety of minimally invasive procedures such as carotid stenting against medical treatment according to clinical routine in this specific patient group. With CARESTAR, a multicentre, prospective, randomised, parallel-grouped open label and blinded safety endpoint study this gap shall be closed. Given the considerations outlined above, symptomatic non-stenotic carotid disease (SyNC) <50% with neurological symptoms represents a desperate situation, where all available options for contribution to the improvement of the patient's state of health or to the prevention of secondary diseases should be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute ischemic stroke or acute retinal artery ischemia within the last two weeks related to symptomatic non-stenotic carotid disease (SyNC) and high-risk carotid plaque features

  * Ipsilateral acute ischemic stroke must be determined by acute ischemic infarct on DWI or CT OR
  * by neurological symptoms indicating ipsilateral cortical deficits consistent with ischemia in the territory of the internal carotid artery and after exclusion of a significant microangiopathy
  * Acute retinal artery ischemia must be determined by ophthalmologic examination
* Patients with no other identifiable cause of stroke, evaluated using standard echocardiographic examinations to exclude cardiogenic or aortogenic sources of embolism
* Symptomatic non-stenotic carotid disease defined as one or more plaques in the ipsilateral internal carotid artery causing 10-49% luminal narrowing AND
* Presence of high-risk plaque features which must be determined through visual inspection on CTA or MRI (Ultrasound findings alone are insufficient; features must be confirmed by CTA or MRI to meet the criteria):

  * Identification of at least two of the following characteristics Plaque thickness ≥ 3mm Irregular plaque surface Ulceration <50% plaque calcification Lipid-rich necrotic core
  * and/or identification of at least one of the following characteristics Intraplaque haemorrhage
* Presence of carotid web characterized as shelf-like/linear, smooth filling defects
* Plaque assessment including evaluation of the presence of high-risk features by routine imaging (CTA, MRI) confirmed by an independent CoreLab
* Signed Informed Consent Form
* Patient ≥ 18 years
* mRS ≤ 3 at time of randomisation
* Dual antiplatelet therapy (DAPT) according to standard of care before endovascular treatment

Exclusion Criteria:

* Patients with acute complete occlusion of the carotid artery in an emergency setting
* Incidence of acute infarcts in other vascular (i.e., not ipsilateral carotid) territories
* Patients in whom the stroke was likely caused by one of the following diseases:
* Small vessel disease

  * Large vessel atherosclerotic disease ≥ 50%
  * Cardioembolism
  * Other known disease e.g. vasculitis
* Predominantly calcified Plaques (≥50% calcified plaque components on CT-Angio)
* Patients presenting with intraluminal carotid thrombus (e.g. characterized by 'donut sign' on CTA)
* Patients with highly tortuous vessels (>90°) which may prevent access or safe insertion of the stent
* Patients with post-CEA re-stenosis or post-CAS re-stenosis
* Patients with blood coagulation disorders
* Patients in whom access to the carotid lesion is impossible or associated with an increased risk of procedural complications
* Patients with lesions in the ostium of the common carotid artery
* Patients with known hypersensitivity to nickel-titanium
* Patients who are allergic to heparin
* Any known conditions that affect life expectancy to less than 12 months
* Any known conditions associated with an increased risk of endovascular treatment
* Patients not able to visit the outpatient clinic for annual follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with <50% symptomatic non-stenotic carotid disease (SyNC) who were treated after randomisation by:
  Endovascular Treatment Group: Stenting + medical management
  o This group will be both given medical treatment according to standard clinical routine and treated by carotid artery stenting with the high coverage carotid stent (CARESTO® heal, Acandis® Pforzheim)
  Best medical treatment group: Medical management alone
  o This group will be given medical treatment according to standard clinical routine
Sampling Method: Probability Sample
Enrollment: 536 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2031-10-31 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint as rate of events of ipsilateral recurrent ischemic stroke or ipsilateral retinal artery ischemia analysed as time to first occurence | Through study completion, an average of 54 months
  Ipsilateral recurrent ischemic stroke or ipsilateral retinal artery ischemia during follow-up analysed as time to first occurence

SECONDARY OUTCOMES:
Secondary Endpoint of Incidence of events and change from functional status | Through study completion, an average of 54 months
  * Each of the components of the primary outcome: Rate of Ipsilateral recurrent ischemic stroke or ipsilateral retinal artery ischemia
  * A composite of rate of ipsilateral recurrent ischemic stroke or ipsilateral retinal artery ischemia during follow-up or any symptomatic stroke, death, or myocardial infarction within 30 ± 10 days after randomisation
  * A composite of rate of disabling ipsilateral recurrent ischemic stroke or ipsilateral retinal artery ischemia during follow-up or disabling stroke, death, or disabling myocardial infarction within 30 ± 10 days after randomisation, where disabling is defined as any event resulting in a worsening by at least one point on the modified Rankin Scale (mRS) (e.g. 0-6)
  * Rate of any change in functional status from admission to follow-up visits, assessed using the Canadian Outcome Scale for MinOr Stroke (COSMOS), comparing post-stroke functioning at follow-up to the patient's functional status recorded at hospital admission (e.g. 0-6)
Secondary Endpoint of Incidence of events and change from functional status | Through study completion, an average of 54 months
  * Occurrence of stroke between randomisation and treatment initiation for both groups
  * Occurrence of further complications during follow-up:
    * Rate of any stroke (ischemic or haemorrhagic) as time to the first occurrence
    * Rate of death (any) as time to event endpoint
    * Rate of transient ischemic attack (TIA) as time to the first occurrence
    * Rate of ipsilateral transient ocular symptoms, e.g., Amaurosis fugax, as time to the first occurrence
    * Rate pf myocardial infarction as time to the first occurrence
    * Rate of device- and procedure-related (S)AEs
    * Rate of plaque progression or re-stenosis requiring (further) treatment (e.g., carotid artery stenting, carotid endarterectomy)
    * Change in the modified Rankin Scale (mRS) score at 30±10 days and during annual status checks at 12-72 months, as compared to mRS pre-randomisation (Delta mRS) (e.g. mRS 0-6)

OTHER OUTCOMES:
Safety Endpoint as rate of symptomatic stroke, death, or myocardial infarktion as safety endpoint | 30 ± 10 days after randomisation
  Any symptomatic stroke, death, or myocardial infarction within 30 ± 10 days after randomisation, evaluated through blinded functional assessment based on in-hospital follow-up and/or telephone interviews with statistical comparison of the endovascular treatment arm to a performance goal derived from the best available evidence in previous stenting studies
Treatment Endpoints as rate of (Peri-)procedural complications | Periprocedural
  •(Peri-)procedural complications related to endovascular treatment, assessed up to in-hospital follow-up/discharge and based on clinical routine measurements
  * Examination of functional status (mRS - e.g. 0-6) and neurological status (NIHSS e.g. Number)
  * Symptomatic intracranial haemorrhage (SICH) defined as any intracranial haemorrhage causing any clinical deterioration and/or SICH as defined in SITS-MOST: Local or remote parenchymal hematoma type 2 on the imaging scan, plus neurological deterioration, as indicated by a score on the NIHSS ≥ 4 points, or leading to death
  * Lumen narrowing post-stent placement per NASCET criteria (%)
  * Major bleeding defined as occurring when at least one of the following conditions is met:
  * Fatal bleeding
  * Symptomatic bleeding in a critical organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, or intramuscular bleeding associated with compartment syndrome.
  * A hemoglobin drop of ≥2 g/dL.
Exploratory outcomes as rate of morphological changes | Through study completion, an average of 54 months
  •Rate of morphological changes observed in high-risk plaques due to their progression and potential implications for patient management strategies at annual follow-up related to ultrasound examination

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Complicated Carotid Artery Plaques as a Cause of Cryptogenic Stroke — https://pubmed.ncbi.nlm.nih.gov/33153580/